CLINICAL TRIAL: NCT02524873
Title: Assessment of the Relationship Between Genes That Encode Proteins Important in Blood Pressure Regulation and Blood Pressure Therapy in Patients With Hypertension
Brief Title: Relationship Between Genes Important in Blood Pressure Regulation and Blood Pressure Therapy in Hypertension
Status: Completed | Type: Observational
Sponsor: Geneticure, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GTC01
Record Dates: First submitted 2015-08-10; First posted 2015-08-17 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Geneticure Collection Kit for Pharmaocogenetics of Hypertension — Buccal (cheek) swab kit for DNA collection for analysis of genes for hypertension

SUMMARY:
Whether patients with a functional genotype of a protein important in blood pressure regulation respond better to a drug therapy class/combination of therapy classes that target that specific pathway using the Geneticure panel for high blood pressure

DETAILED DESCRIPTION:
2.1 Study Design and Protocol Overview This is a post-hoc association study of patients who have been diagnosed with high blood pressure and have been stable on medication treatment for at least 6 months. The purpose of this study is to evaluate the relationship between optimal medication therapy (or the therapy that has resulted in the most stable blood pressure for that particular patient) and the predicted optimal medication therapy based on a patient's genetic profile.

Chart reviews for the patient's history of antihypertensive therapy will be coupled with buccal swabs and blood pressure readings collected from eligible patients who have provided informed consent. The swab will be analyzed for fourteen genetic variants that are associated with antihypertensive therapy response (efficacy, side-effects).

2.2 Study Objective To assess the relationship between the drug therapy class/combination of therapy classes that resulted in the best blood pressure control for a patient vs. what the Geneticure high blood pressure panel would have predicted.

2.3 Secondary Objectives

* To assess the clinical time to achieve optimal blood pressure treatment.
* To assess the number of office visits required to achieve optimal blood pressure treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to provide informed consent
2. Subject is ≥ 30 and ≤ 70 years of age
3. Subject with diagnosis of Hypertension for a minimum of 1 year
4. Subject has been on the same class/classes of blood pressure medication for a minimum of 6 months. Note: A change in dosage, frequency, or specific medication is acceptable as long as there have been no changes to the class/classes of medications prescribed.
5. Subject with a Body Mass Index (BMI) ≥ 19 and ≤ 35
6. Subject is currently prescribed and taking one of the following classes of medications alone or in combination with each other or a Ca+ channel blocker.

   * Diuretics
   * ACE Inhibitors
   * Angiotensin Receptor Blocker (ARB)
   * Beta-blockers

Exclusion Criteria:

1. Subject has clinically significant kidney disease as determined by the investigator.
2. Subject has clinically significant cardiac disease as determined by the investigator.
3. Subject has clinically significant vascular disease as determined by the investigator.
4. Subject has a diagnosis of secondary hypertension or is experiencing a complication of pregnancy.
5. Subject is currently prescribed and taking any additional class of medication(s) for high blood pressure not included in the list above, with the exception of a Ca+ channel blocker.
6. Subject has Systolic BP > 190 or Diastolic BP > 120 documented within the six months prior to visit.
7. Subject has a regular alcohol intake of greater than 21 units per week in the past 6 months
8. Subject has smoked greater than two packs of cigarettes (total) or equivalent nicotine intake in the past 6 months.
9. Subject has an anticipated survival less than 12 months.
10. Any other reason that the subject is inappropriate for study enrollment in the opinion of the Investigator.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure changes (using sphygmomanometry) in response to therapy according to genes important in blood pressure regulation | one year
  To assess the relationship between the drug therapy class/combination of therapy classes that resulted in the best blood pressure control for a patient vs. what the Geneticure high blood pressure panel would have predicted. We will assess blood pressure values (systolic and diastolic blood pressure, in mmHg) at rest in patients on different blood pressure medications.

SECONDARY OUTCOMES:
The clinical time to achieve optimal blood pressure treatment | One year
The number of office visits required to achieve optimal blood pressure treatment. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Krista Kleve, Study Director — RCRI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johnson MW, Sprissler R, Olson TP, Beenken GW, Snyder EM. Multi-Gene Pharmacogenetics and Blood Pressure Control in Patients with Hypertension. The FASEB Journal 30:942.1. 2016
- [Result] Johnson MW, Sprissler R, Olson TP, Beenken GW, Snyder EM. Time to Blood Pressure Control According to Drug Class in Patients with Hypertension. The FASEB Journal 30:941.12. 2016.